CLINICAL TRIAL: NCT03364842
Title: Furosemide: Would it Help to Improve the Lungs During Aortic Coarctation Surgery
Brief Title: Furosemide and Coarctation Surgery Lung Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kareem, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fuurosemide and coarctation
Record Dates: First submitted 2017-11-21; First posted 2017-12-07 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Complication
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- F group (Experimental): Furosemide group
  Interventions: Drug: Furosemide
- C group (No Intervention): Control group

INTERVENTIONS:
Drug: Furosemide — Administering furosemide
  Arms: F group

SUMMARY:
in our study the investigators give furosemide during surgery for repair of aortic coarctation via lateral thoracotomy and evaluated lung complications in comparison to control group

ELIGIBILITY:
Inclusion Criteria:

* coarctation of aorta

Exclusion Criteria:

* heart failure, bleeding diathesis, associated cardiac congenital anomalies

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
lung ultrasonography scale > 24 | a 1 year study

SECONDARY OUTCOMES:
Pao2/ Fio2 ratio | a 1 year study

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided